CLINICAL TRIAL: NCT00907868
Title: A Multicentric Phase III Trial Evaluating the Impact of a Radiation Boost (16Gy) After Breast Conserving Surgery and a Whole Breast Irradiation (50Gy) for DCIS
Brief Title: Breast-Conserving Surgery and Whole-Breast Radiation Therapy With or Without Additional Radiation Therapy to the Tumor in Treating Women With Ductal Carcinoma in Situ (BONBIS)
Acronym: BONBIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000636007; RECF0911 (Registry Identifier: INCA); VA-2008/25 (Other: Organization protocol ID); 2008-A00494-51 (Other: ID-RCB number)
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Active Comparator): Patients undergo whole breast irradiation (WBI) once daily for 5 weeks (weekdays only).
  Interventions: Radiation: whole breast irradiation
- Arm II (Experimental): Patients undergo WBI as in arm I and a radiation tumor bed boost once daily for 8 days (weekdays only).
  Interventions: Radiation: partial breast irradiation; Radiation: whole breast irradiation

INTERVENTIONS:
Radiation: partial breast irradiation — Patients undergo radiation tumor bed boost
  Arms: Arm II
Radiation: whole breast irradiation — Patients undergo whole breast irradiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether whole-breast radiation therapy is more effective when given with or without additional radiation therapy to the tumor in treating patients with ductal carcinoma in situ.

PURPOSE: This randomized phase III trial is studying breast-conserving surgery followed by whole-breast radiation therapy to see how well it works when given with or without additional radiation therapy to the tumor in treating women with ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate and compare local recurrence-free survival of women with ductal breast carcinoma in situ (DCIS) treated with breast-conserving surgery followed by whole breast irradiation with vs without a radiation tumor bed boost.

Secondary

* Compare relapse-free survival between the two arms.
* Compare overall survival.
* Compare acute and late toxicities.
* Compare cosmetic results and quality of life.
* Identify patients at risk for late toxicities using a biological test.

Tertiary

* Store blood samples at the CEPH (French Center of the Human Polymorphism Center) for polymorphism analyses.

OUTLINE: This is a multicenter study. All patients undergo breast-conserving surgery (after a single intervention or second excision) with a margin ≥ 1 mm. A superficial or deep margin is acceptable if the surgery has left the skin tissue or the fascia pectoral muscle, respectively. Twelve weeks later, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo whole breast irradiation (WBI) once daily, 5 days a week for 5 weeks.
* Arm II: Patients undergo WBI as in arm I. Patients also undergo a radiation tumor bed boost once daily for 8 fractions (weekdays only) over 2 weeks.

Quality of life will be assessed.

After completion of study treatment, patients are followed up every 6 months for 5 years and then annually for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ of the breast

  * No invasive component
  * No clinically palpable lymph node or presence of tumor cells in the sentinel lymph node (if done)
  * No local recurrence of a primary breast cancer
  * No multicentric or multifocal tumors not suitable for conservative surgery R0 with a margin ≥ 1 mm
* Has undergone bilateral mammography within 6 months before randomization

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 5 years
* Not pregnant
* Available for long-term follow up
* No history of in situ carcinoma in the contralateral breast
* No history of another cancer except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No uncontrolled cardiac, renal, or pulmonary disease
* No uncontrolled systemic disease (e.g., lupus erythematosus or scleroderma)
* No HIV positivity
* Affiliated with the social health system
* No psychological, familial, sociological, or geographical situations that preclude compliance with study treatment and follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation in another therapeutic trial (participation in epidemiologic studies is allowed)

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence | up to 15 years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: David Azria, MD, PhD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azria D, Gourgou S, Sozzi WJ, Zouhair A, Mirimanoff RO, Kramar A, Lemanski C, Dubois JB, Romieu G, Pelegrin A, Ozsahin M. Concomitant use of tamoxifen with radiotherapy enhances subcutaneous breast fibrosis in hypersensitive patients. Br J Cancer. 2004 Oct 4;91(7):1251-60. doi: 10.1038/sj.bjc.6602146. PMID 15328527
- [Background] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Background] EORTC Breast Cancer Cooperative Group; EORTC Radiotherapy Group; Bijker N, Meijnen P, Peterse JL, Bogaerts J, Van Hoorebeeck I, Julien JP, Gennaro M, Rouanet P, Avril A, Fentiman IS, Bartelink H, Rutgers EJ. Breast-conserving treatment with or without radiotherapy in ductal carcinoma-in-situ: ten-year results of European Organisation for Research and Treatment of Cancer randomized phase III trial 10853--a study by the EORTC Breast Cancer Cooperative Group and EORTC Radiotherapy Group. J Clin Oncol. 2006 Jul 20;24(21):3381-7. doi: 10.1200/JCO.2006.06.1366. Epub 2006 Jun 26. PMID 16801628
- [Background] Bijker N, Peterse JL, Duchateau L, Julien JP, Fentiman IS, Duval C, Di Palma S, Simony-Lafontaine J, de Mascarel I, van de Vijver MJ. Risk factors for recurrence and metastasis after breast-conserving therapy for ductal carcinoma-in-situ: analysis of European Organization for Research and Treatment of Cancer Trial 10853. J Clin Oncol. 2001 Apr 15;19(8):2263-71. doi: 10.1200/JCO.2001.19.8.2263. PMID 11304780
- [Background] Cutuli B, Cohen-Solal-le Nir C, de Lafontan B, Mignotte H, Fichet V, Fay R, Servent V, Giard S, Charra-Brunaud C, Lemanski C, Auvray H, Jacquot S, Charpentier JC. Breast-conserving therapy for ductal carcinoma in situ of the breast: the French Cancer Centers' experience. Int J Radiat Oncol Biol Phys. 2002 Jul 15;53(4):868-79. doi: 10.1016/s0360-3016(02)02834-1. PMID 12095552
- [Background] Cutuli B, Fourquet A, Luporsi E, Arnould L, Caron Y, Cremoux Pd, Dilhuydy JM, Fondrinier E, Fourme E, Giard-Lefevre S, Blanc-Onfroy ML, Lemanski C, Mauriac L, Sigal-Zafrani B, Tardivon A, This P, Tunon de Lara C, Kirova Y, Fabre N; Federation of French Cancer Centres (FNCLCC), et le groupe de travail SOR. [Standards, Options and Recommendations for the management of ductal carcinoma in situ of the breast (DCIS): update 2004]. Bull Cancer. 2005 Feb;92(2):155-68. French. PMID 15749645
- [Background] Emdin SO, Granstrand B, Ringberg A, Sandelin K, Arnesson LG, Nordgren H, Anderson H, Garmo H, Holmberg L, Wallgren A; Swedish Breast Cancer Group. SweDCIS: Radiotherapy after sector resection for ductal carcinoma in situ of the breast. Results of a randomised trial in a population offered mammography screening. Acta Oncol. 2006;45(5):536-43. doi: 10.1080/02841860600681569. PMID 16864166
- [Background] Ernster VL, Barclay J, Kerlikowske K, Grady D, Henderson C. Incidence of and treatment for ductal carcinoma in situ of the breast. JAMA. 1996 Mar 27;275(12):913-8. PMID 8598618
- [Background] Fine JP. Regression modeling of competing crude failure probabilities. Biostatistics. 2001 Mar;2(1):85-97. doi: 10.1093/biostatistics/2.1.85. PMID 12933558
- [Background] Fisher B, Dignam J, Wolmark N, Wickerham DL, Fisher ER, Mamounas E, Smith R, Begovic M, Dimitrov NV, Margolese RG, Kardinal CG, Kavanah MT, Fehrenbacher L, Oishi RH. Tamoxifen in treatment of intraductal breast cancer: National Surgical Adjuvant Breast and Bowel Project B-24 randomised controlled trial. Lancet. 1999 Jun 12;353(9169):1993-2000. doi: 10.1016/S0140-6736(99)05036-9. PMID 10376613
- [Background] Fisher B, Land S, Mamounas E, Dignam J, Fisher ER, Wolmark N. Prevention of invasive breast cancer in women with ductal carcinoma in situ: an update of the National Surgical Adjuvant Breast and Bowel Project experience. Semin Oncol. 2001 Aug;28(4):400-18. doi: 10.1016/s0093-7754(01)90133-2. PMID 11498833
- [Background] Gagliardi G, Lax I, Soderstrom S, Gyenes G, Rutqvist LE. Prediction of excess risk of long-term cardiac mortality after radiotherapy of stage I breast cancer. Radiother Oncol. 1998 Jan;46(1):63-71. doi: 10.1016/s0167-8140(97)00167-9. PMID 9488129
- [Background] Ho AY, Atencio DP, Peters S, Stock RG, Formenti SC, Cesaretti JA, Green S, Haffty B, Drumea K, Leitzin L, Kuten A, Azria D, Ozsahin M, Overgaard J, Andreassen CN, Trop CS, Park J, Rosenstein BS. Genetic predictors of adverse radiotherapy effects: the Gene-PARE project. Int J Radiat Oncol Biol Phys. 2006 Jul 1;65(3):646-55. doi: 10.1016/j.ijrobp.2006.03.006. PMID 16751059
- [Background] Houghton J, George WD, Cuzick J, Duggan C, Fentiman IS, Spittle M; UK Coordinating Committee on Cancer Research; Ductal Carcinoma in situ Working Party; DCIS trialists in the UK, Australia, and New Zealand. Radiotherapy and tamoxifen in women with completely excised ductal carcinoma in situ of the breast in the UK, Australia, and New Zealand: randomised controlled trial. Lancet. 2003 Jul 12;362(9378):95-102. doi: 10.1016/s0140-6736(03)13859-7. PMID 12867108
- [Background] Omlin A, Amichetti M, Azria D, Cole BF, Fourneret P, Poortmans P, Naehrig D, Miller RC, Krengli M, Gutierrez Miguelez C, Morgan D, Goldberg H, Scandolaro L, Gastelblum P, Ozsahin M, Dohr D, Christie D, Oppitz U, Abacioglu U, Gruber G. Boost radiotherapy in young women with ductal carcinoma in situ: a multicentre, retrospective study of the Rare Cancer Network. Lancet Oncol. 2006 Aug;7(8):652-6. doi: 10.1016/S1470-2045(06)70765-3. PMID 16887482
- [Background] Ozsahin M, Crompton NE, Gourgou S, Kramar A, Li L, Shi Y, Sozzi WJ, Zouhair A, Mirimanoff RO, Azria D. CD4 and CD8 T-lymphocyte apoptosis can predict radiation-induced late toxicity: a prospective study in 399 patients. Clin Cancer Res. 2005 Oct 15;11(20):7426-33. doi: 10.1158/1078-0432.CCR-04-2634. PMID 16243816
- [Background] Solin LJ, Fourquet A, Vicini FA, Haffty B, Taylor M, McCormick B, McNeese M, Pierce LJ, Landmann C, Olivotto IA, Borger J, Kim J, de la Rochefordiere A, Schultz DJ. Mammographically detected ductal carcinoma in situ of the breast treated with breast-conserving surgery and definitive breast irradiation: long-term outcome and prognostic significance of patient age and margin status. Int J Radiat Oncol Biol Phys. 2001 Jul 15;50(4):991-1002. doi: 10.1016/s0360-3016(01)01517-6. PMID 11429227
- [Result] Bourgier C, Cowen D, Castan F, Lemanski C, Gourgou S, Rivera S, Labib A, Peignaux K, Blanc-Onfroy ML, Benyoucef A, Mege A, Douadi-Gaci Z, Racadot S, Latorzeff I, Schick U, Jacquot S, Massabeau C, Guilbert P, Geffrelot J, Ellis S, Lecouillard I, Breton-Callu C, Richard-Tallet A, Boulbair F, Cretin J, Belkacemi Y, Bons F, Azria D, Fenoglietto P. Quality assurance program and early toxicities in the phase III BONBIS randomized trial evaluating the role of a localized radiation boost in ductal carcinoma in situ. Radiother Oncol. 2021 Nov;164:57-65. doi: 10.1016/j.radonc.2021.09.014. Epub 2021 Sep 24. PMID 34571090
- [Result] Bourgier C, Mollevi C, Cowen D, Castan F, Lemanski C, Gourgou S, Rivera S, Labib A, Peignaux K, Blanc-Onfroy ML, Benyoucef A, Mege A, Douadi-Gaci Z, Racadot S, Latorzeff I, Schick U, Jacquot S, Massabeau C, Guilbert P, Geffrelot J, Ellis S, Lecouillard I, Breton-Callu C, Richard-Tallet A, Boulbair F, Belliere A, Magne N, Belkacemi Y, Bons F, Fenoglietto P, Azria D. Late Toxicities and Quality of Life After a Radiation Boost for Breast Ductal Carcinoma In Situ: Boost or No Boost in DCIS Randomized Trial. Int J Radiat Oncol Biol Phys. 2026 Jan 1;124(1):109-121. doi: 10.1016/j.ijrobp.2025.07.1442. Epub 2025 Jul 31. PMID 40752655
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.e-cancer.fr/Professionnels-de-sante/Le-registre-des-essais-cliniques/Le-registre-des-essais-cliniques/Etudes-cliniques/BONBIS-Essai-de-phase-3-randomise-evaluant-l-efficacite-d-un-complement-de-radiotherapie-apres-traitement-conservateur-chez-des-patientes-ayant-un-cancer-du-sein.-essai-clos-aux-inclusions